CLINICAL TRIAL: NCT05584007
Title: A Blinded, Non-inferiority Phase III Trial of 5 Versus 7 Days of Oral Flucloxacillin in Primary Care Patients With Lower Limb Cellulitis
Brief Title: Cellulitis Optimal Antibiotic Treatment
Acronym: COAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University of East Anglia (Other); University of Nottingham (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERGO 67073
Record Dates: First submitted 2022-09-07; First posted 2022-10-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cellulitis of Leg
Keywords: Primary care; Antibiotic treatment; Antibiotic resistance; Pain; Cost consequences
MeSH Terms: conditions — Pain | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: A phase III blinded, multi-center, non-inferiority trial assessing the effectiveness and safety of 5 days vs 7 days of oral flucloxacillin 500mg QDS for lower leg cellulitis, and to evaluate the cost-consequences of a shorter course from an NHS and personal perspective. Participants will be recruited in NHS primary care settings in England and Wales. We will primarily recruit through general practices but will explore the possibility of recruiting through out-of-the-hours and urgent care settings.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To facilitate ease of recruitment and avoid treatment delay, participants will be provided with an NHS prescription for flucloxacillin 500mg QDS for the first 5 days. A blinded medication pack will be sent by next day delivery, containing flucloxacillin 500mg QDS, or matched placebo QDS for the final 2 days. Participants will be informed that the capsules in this pack may look different from the capsules they were taking on days 1-5. Participants experiencing significant clinical deterioration, as judged by their clinician, may have their antibiotic treatment changed or be prescribed additional antibiotic courses. Any changes or additional use of antibiotics will be recorded, and the patient and clinician will remain blinded unless unblinding is deemed necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Placebo Comparator): Flucloxacillin 500mg four times a day (QDS) for 5 days (unblinded NHS prescription) followed by blinded placebo QDS for 2 days (5 days of antibiotic)
  Interventions: Drug: Flucloxacillin Only Product in Oral Dose Form; Drug: Placebo Only Product in Oral Dose Form
- Control (Active Comparator): Flucloxacillin 500mg QDS for 5 days (unblinded NHS prescription) followed by flucloxacillin 500mg QDS (blinded) for 2 days (7 days of antibiotic)
  Interventions: Drug: Flucloxacillin Only Product in Oral Dose Form

INTERVENTIONS:
Drug: Flucloxacillin Only Product in Oral Dose Form — Patients will be prescribed flucloxacillin 500mg QDS for 5 days followed by blinded flucloxacillin 500mg for 2 days, reaching a total of 7 days of antibiotic treatment
Drug: Placebo Only Product in Oral Dose Form — Patients will be prescribed flucloxacillin 500mg QDS for 5 days followed by a blinded placebo for 2 days, reaching a total of 5 days of antibiotic treatment
  Arms: Intervention

SUMMARY:
To determine whether a short course of oral flucloxacillin (5 days) is non-inferior to a standard course (7 days) in terms of pain over days 6-14 (indicative of persistence or recurrence associated with the symptoms of most importance to patients) in adults with cellulitis of the leg presenting in primary care.

DETAILED DESCRIPTION:
Cellulitis is a deep infection of the skin and subcutaneous tissues and most often occurs in the legs. It is a painful condition that is associated with inflammation and swelling of the site, and often systemic symptoms such as fever, headache, muscle aches, malaise, and fatigue. Patients report feeling unwell and that it has a significant impact on their mobility and ability to carry out their usual activities. NICE guidelines recommend oral flucloxacillin 500-1000 mg four times daily for 5-7 days as first-line treatment for most patients with cellulitis in the community, but most prescriptions are dispensed for a 7-day course. We will be assessing the effectiveness and safety of a 5-day treatment vs. the standard 7-day treatment. We also aim to evaluate the cost-consequences of a shorter course from an NHS and personal perspective. Participants will be randomly allocated to one of two groups. In addition to usual care, participants will either be assigned to a 5-day oral flucloxacillin course or a standard 7-day flucloxacillin course. Participants will be prescribed a 5-day course of oral flucloxacillin, and two additional tablets will be posted to the participants which will either be the antibiotic or a placebo tablet. Participants will be asked to fill out daily questionnaires and express their experiences with the shortened course and taking part in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 years or older
* Currently showing symptoms of cellulitis (such as pain, tenderness, redness, other change in skin color, warmth to touch) in one leg for 10 days or less
* Pain rated as 3/10 or higher on a numerical rating scale (0-10) at baseline assessment
* Be willing to be randomized to either trial arm (5-day or 7-day treatment)
* Able to complete trial procedures in the English language.

Exclusion Criteria:

* Have penicillin allergy
* Have bilateral cellulitis
* Have had antibiotics for cellulitis within the past month
* Have post-operative cellulitis (within 30 days of operative procedures on the same leg)
* Have cellulitis resulting from human/animal bite injury
* Have Cellulitis associated with chronic (>6 weeks) leg ulceration
* Require immediate hospital admission or out-patient intravenous antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | Days 7-16
  Self-reported pain (measured using the Pain Numeric Rating Scale (0-10))

SECONDARY OUTCOMES:
Use of additional antibiotics | Up to day 28
  Any reported use of antibiotics other than the initial 5 days of flucloxacillin and 2 days of IMP)
Patient-reported assessment of how well they are feeling | Days 6-14
  Numeric rating scale NRS (0-10) and assessed as repeated measures
Health related quality of life | Days 6-14
  EQ-5D-5L - values, and individual dimension (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) level scores using repeated measures.
Health related quality of life used to estimate Quality Adjusted- Life Years (QALYs) | Days 6-14
  EQ-5D-5L - values, and individual dimension (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) level scores using repeated measures.
Leg swelling and warmth | Day 7, 14, 21, 28
  Participant reported questionnaire
Time until self-reported recovery | Day 7, 14, 21, 28
  Participant reported questionnaire
Time until self-assessed extent of cellulitis starts to reduce (with no subsequent increase) | Day 7, 14, 21, 28
  Participant reported questionnaire
Hospital admissions | 12 months
  Number of hosptial admissions since randomisation, collected from primary care notes review
Recurrent cellulitis episodes over 12 months (number of episodes) | 12 months
  Recurrent cellulitis episodes over 12 months (number of episodes) since randomisation, collected from primary care notes review
Complications over 12 months | 12 months
  Number of reported complications since randomisation, collected from primary care notes review

CONTACTS AND LOCATIONS:
Locations (1):
- Royal South Hants Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data from all centers will be analyzed together and published as soon as possible.
  Planned publication of the results in a high-impact peer-reviewed journal. Planned publication of protocol in a peer-review journal. The datasets generated and/or analyzed during the current study will be published as a supplement to the publication of the results. Individual investigators may not publish data concerning their patients that are directly relevant to questions posed by the trial until the Trial Management Group (TMG) has published its report. The TMG will form the basis of the Writing Committee and advise on the nature of publications.